CLINICAL TRIAL: NCT03139084
Title: An Observational, Non-interventional, Multicenter Study to Evaluate the Efficacy and Safety of Upfront Combination of Bosentan and Tadalafil in Pulmonary Arterial Hypertension in Greek Patients
Brief Title: Efficacy and Safety of Upfront Combination of ΒΟsentan and ΤΑdalafil in Pulmonary Arterial Hypertension
Acronym: BOTA-PAH
Status: Withdrawn | Type: Observational
Why Stopped: Updated results by guidelines and bibliography
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017-BSN-EL-73
Record Dates: First submitted 2017-04-28; First posted 2017-05-03 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The development of disease-targeted drugs for the treatment of pulmonary arterial hypertension (PAH) has significantly improved within the last years. Combining drug products with different mechanisms of action such as Endothelin-Receptor-Antagonists (ERAs) and Phosphodiesterase-Type-5-inhibitors (PDE-5-Inhibitors) has become increasingly important for the treatment of PAH. Recently, the results of the AMBITION study reported that an upfront combination treatment of ambrisentan and tadalafil immediately after diagnosis leads to a delayed disease progression. On the other hand, the sequential combination of bosentan and sildenafil did not show a similar positive clinical effect and this was attributed to a negative clinically relevant pharmacodynamic drug-drug interaction. Although, recent guidelines have extrapolated that initial upfront combination treatment follows a class effect in terms of efficacy and safety, there is an imperative need to support this notion with other combinations of ERAs and PDE-5-Inhibitors.

DETAILED DESCRIPTION:
The primary objective of BOTA study is to compare the change in clinical and hemodynamic measures of PAH after the initiation of first line combination therapy with bosentan and tadalafil in adult patients with PAH. The safety and tolerability of first line combination therapy will also be evaluated.

In patients with PAH initial upfront combination treatment with bosentan and tadalafil

1. Improves

   * Exercise capacity as expressed by distance walked in six minute walk test and WHO functional class
   * Hemodynamics in terms of pulmonary vascular resistance (PVR), mean pulmonary artery pressure (mPAP) reduction and cardiac index (CI) elevation
   * Quality of life
   * NTproBNP serum levels
   * Echocardiographic prognostic parameters such as right atrial area and presence of pericardial effusion.
2. Is safe as assessed by

   * Liver function markers such as serum SGOT and SGPT levels
   * Hemoglobin levels

ELIGIBILITY:
Inclusion Criteria:

Male or females between 18 to 75 years of age at inclusion

Diagnosis of PAH due to the following:

* Idiopathic Primary Pulmonary Arterial Hypertension (IPAH)
* Hereditary PAH
* PAH secondary to connective tissue disease
* PAH diagnosis confirmed by right heart catheterization performed within 3 months prior to study enrolment Subjects must weigh at least 40 kg at inclusion Subject must have a current diagnosis of being in World Health Organisation (WHO) Functional Class II or III.

Treatment PAH naïve subjects PAH documented by

* mPAP ≥25mmHg,
* pulmonary capillary wedge pressure (PCWP) or
* left ventricular end-diastolic pressure (LVEDP) ≤15mmHg and
* PVR ≥3 Wood Units. Subject must walk a distance of ≥125m and ≤500m at the screening visit

Exclusion Criteria:

* History of pulmonary embolism
* No prior treatment with PDE-5 inhibitors
* History of chronic lung disease / restrictive lung disease (eg, chronic obstructive pulmonary disease (COPD) or scleroderma) with impairment of lung function
* Current treatment with nitrates or nitric oxide
* Significant (ie, >2+) valvular disease other than tricuspid regurgitation or pulmonary regurgitation
* History of cardiac arrest, respiratory arrest, hemodynamic collapse, CPR, ventricular tachycardia, ventricular fibrillation, or uncontrolled atrial fibrillation

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed patients with PAH
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in the N-Terminal Pro-B-Type Natriuretic Peptide at Month 6 | 6 months
  N-Terminal Pro-B-Type Natriuretic Peptide (NT-proBNP) is a surrogate marker of heart failure. The geometric mean ratio will be calculated as the ratio between the month 6 value and the Baseline value and presented as percent change = 100 * (geometric mean ratio - 1). The Baseline value is the last value prior to administration of study drug; this may be prior to or on the day of study drug initiation.

SECONDARY OUTCOMES:
Number of Participants With First Adjudicated Clinical Failure (CF) Event | 6 months
  Hospitalisation for Worsening PAH, Disease Progression, Unsatisfactory Clinical Response
Time to first clinical worsening (TTCW) event | 6 months
  TTCW defined as the number of days between first dose of study drug and the occurrence of a predefined clinical worsening event.
Percentage of Participants With a Satisfactory Clinical Response at Month 6 | 6 months
  A satisfactory clinical response at month 6 is defined as a participant who meets all of the following criteria: 10% improvement in 6MWD compared with Baseline;
Change From Baseline in the World Health Organization Functional Class at month 6 | 6 months
  Change From Baseline in the World Health Organization Functional Class Time Frame: Baseline and Month 6 The WHO Functional Class (FC) indicates the severity of PAH and is an adaptation of the New York Heart Association classification.
Change From Baseline in the 6 Minute Walk Distance (6MWD) Test at month 6 | 6 months
  Change From Baseline in the 6 Minute Walk Distance (6MWD) Test at month 6
  MWD is the distance a participant can walk in 6 minutes. The 6-minute walk distance (6MWD) test measures the distance that a participant can walk in a period of 6 minutes.
Change From Baseline in Borg Dyspnea Index at month 6 | 6 months
  Borg Dyspnea Index (BDI) indicates the degree of breathlessness after completion of the 6 minute walk test.
Quality of Life | 6 moths
  Change in emPHasis-10 questionnaire score

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Galie N, Barbera JA, Frost AE, Ghofrani HA, Hoeper MM, McLaughlin VV, Peacock AJ, Simonneau G, Vachiery JL, Grunig E, Oudiz RJ, Vonk-Noordegraaf A, White RJ, Blair C, Gillies H, Miller KL, Harris JH, Langley J, Rubin LJ; AMBITION Investigators. Initial Use of Ambrisentan plus Tadalafil in Pulmonary Arterial Hypertension. N Engl J Med. 2015 Aug 27;373(9):834-44. doi: 10.1056/NEJMoa1413687. PMID 26308684
- [Result] McLaughlin V, Channick RN, Ghofrani HA, Lemarie JC, Naeije R, Packer M, Souza R, Tapson VF, Tolson J, Al Hiti H, Meyer G, Hoeper MM. Bosentan added to sildenafil therapy in patients with pulmonary arterial hypertension. Eur Respir J. 2015 Aug;46(2):405-13. doi: 10.1183/13993003.02044-2014. Epub 2015 Jun 25. PMID 26113687
- [Result] Galie N, Humbert M, Vachiery JL, Gibbs S, Lang I, Torbicki A, Simonneau G, Peacock A, Vonk Noordegraaf A, Beghetti M, Ghofrani A, Gomez Sanchez MA, Hansmann G, Klepetko W, Lancellotti P, Matucci M, McDonagh T, Pierard LA, Trindade PT, Zompatori M, Hoeper M; ESC Scientific Document Group. 2015 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension: The Joint Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of the European Society of Cardiology (ESC) and the European Respiratory Society (ERS): Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC), International Society for Heart and Lung Transplantation (ISHLT). Eur Heart J. 2016 Jan 1;37(1):67-119. doi: 10.1093/eurheartj/ehv317. Epub 2015 Aug 29. No abstract available. PMID 26320113